CLINICAL TRIAL: NCT04986215
Title: Research on the Value of Genomics Research Based on Ultrasound Endoscopic Biopsy in the Differential Diagnosis and Prognostic Evaluation of Pancreatic Occupancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, Associate Professor, Changhai Hospital
Other Study IDs: 2021-PC-Maker(V1.1）
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Space Occupying

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign pancreatic space occupying group
- Malignant pancreatic space occupying group

SUMMARY:
To clarify the value of genomic testing in the clinical diagnosis or prognosis of pancreatic space occupation, provide a basis for the selection of clinical diagnosis methods for pancreatic space occupation, optimize clinical management strategies, and improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85, no gender limit
2. Imaging examinations suggest that the clear pancreas has clear space-occupying lesions
3. Admitted to our department, ready to undergo endoscopic ultrasound biopsy to confirm the diagnosis

Exclusion Criteria:

1. There are contraindications for endoscopic ultrasound biopsy
2. Failed to join the group or refused follow-up due to various reasons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Occupying lesions of the pancreas, specifically including benign diseases and malignant diseases, mainly pancreatic cancer has a very high incidence. Elderly patients, especially those who drink alcohol all year round, have a lot of occurrences, and many patients are already in the middle or advanced stage when they are diagnosed.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Differential microRNA detected by sequencing | June 2023
  The diagnosis of microRNA in pancreatic space occupying
Differential mRNA detected by sequencing | June 2023
  The diagnosis of mRNA in pancreatic space occupying
Differential lncRNA detected by sequencing | June 2023
  The diagnosis of lncRNA in pancreatic space occupying

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Sep 11;371(11):1039-49. doi: 10.1056/NEJMra1404198. No abstract available. PMID 25207767
- [Background] Ilic M, Ilic I. Epidemiology of pancreatic cancer. World J Gastroenterol. 2016 Nov 28;22(44):9694-9705. doi: 10.3748/wjg.v22.i44.9694. PMID 27956793
- [Background] Lin QJ, Yang F, Jin C, Fu DL. Current status and progress of pancreatic cancer in China. World J Gastroenterol. 2015 Jul 14;21(26):7988-8003. doi: 10.3748/wjg.v21.i26.7988. PMID 26185370
- [Background] Gleeson FC, Kipp BR, Caudill JL, Clain JE, Clayton AC, Halling KC, Henry MR, Rajan E, Topazian MD, Wang KK, Wiersema MJ, Zhang J, Levy MJ. False positive endoscopic ultrasound fine needle aspiration cytology: incidence and risk factors. Gut. 2010 May;59(5):586-93. doi: 10.1136/gut.2009.187765. PMID 20427392
- [Background] Erickson RA. EUS-guided FNA. Gastrointest Endosc. 2004 Aug;60(2):267-79. doi: 10.1016/s0016-5107(04)01529-9. No abstract available. PMID 15278063
- [Background] Chu LC, Goggins MG, Fishman EK. Diagnosis and Detection of Pancreatic Cancer. Cancer J. 2017 Nov/Dec;23(6):333-342. doi: 10.1097/PPO.0000000000000290. PMID 29189329
- [Background] He M, Wu C, Xu J, Guo H, Yang H, Zhang X, Sun J, Yu D, Zhou L, Peng T, He Y, Gao Y, Yuan J, Deng Q, Dai X, Tan A, Feng Y, Zhang H, Min X, Yang X, Zhu J, Zhai K, Chang J, Qin X, Tan W, Hu Y, Lang M, Tao S, Li Y, Li Y, Feng J, Li D, Kim ST, Zhang S, Zhang H, Zheng SL, Gui L, Wang Y, Wei S, Wang F, Fang W, Liang Y, Zhai Y, Chen W, Miao X, Zhou G, Hu FB, Lin D, Mo Z, Wu T. A genome wide association study of genetic loci that influence tumour biomarkers cancer antigen 19-9, carcinoembryonic antigen and alpha fetoprotein and their associations with cancer risk. Gut. 2014 Jan;63(1):143-51. doi: 10.1136/gutjnl-2012-303434. Epub 2013 Jan 7. PMID 23300138
- [Background] Cai Q, Zhu C, Yuan Y, Feng Q, Feng Y, Hao Y, Li J, Zhang K, Ye G, Ye L, Lv N, Zhang S, Liu C, Li M, Liu Q, Li R, Pan J, Yang X, Zhu X, Li Y, Lao B, Ling A, Chen H, Li X, Xu P, Zhou J, Liu B, Du Z, Du Y, Li Z; Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA). Development and validation of a prediction rule for estimating gastric cancer risk in the Chinese high-risk population: a nationwide multicentre study. Gut. 2019 Sep;68(9):1576-1587. doi: 10.1136/gutjnl-2018-317556. Epub 2019 Mar 29. PMID 30926654
- [Background] Nishiwada S, Sho M, Banwait JK, Yamamura K, Akahori T, Nakamura K, Baba H, Goel A. A MicroRNA Signature Identifies Pancreatic Ductal Adenocarcinoma Patients at Risk for Lymph Node Metastases. Gastroenterology. 2020 Aug;159(2):562-574. doi: 10.1053/j.gastro.2020.04.057. Epub 2020 May 4. PMID 32376411
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30207593/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21620466/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25207767/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27956793/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26185370/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20427392/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15278063/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29189329/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23300138/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30926654/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32376411/